CLINICAL TRIAL: NCT04634552
Title: A Phase 1/2, First-in-Human, Open-Label, Dose Escalation Study of Talquetamab, a Humanized GPRC5D x CD3 Bispecific Antibody, in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Talquetamab in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: MonumenTAL-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108920; TALMMY1001-PT3 (Other: Janssen Research & Development, LLC); 2017-002400-26 (EudraCT Number); 2023-504581-29-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05757973 (Approved for marketing)
Record Dates: First submitted 2020-11-16; First posted 2020-11-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hematological Malignancies
Keywords: Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma | interventions — talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 3: Cohort A (Talquetamab) (Experimental): Cohort A will enroll participants with multiple myeloma who have previously received greater than or equal to (>=) 3 prior lines of therapy and have not been exposed to T cell redirection therapies. Participants will receive talquetamab subcutaneously (SC) at a recommended Phase 2 dose (RP2D) selected after review of safety, efficacy, PK, and pharmacodynamic data from Part 1 and Part 2 of this study. All participants (ongoing and those who are in follow-up) will transition to open-label extension (OLE) phase and will continue to receive the study treatment. Upon approval of amendment 19 and notification from the sponsor, participants will transition to the long-term extension (LTE) and will continue to receive study treatment.
  Interventions: Drug: Talquetamab
- Part 3: Cohort B (Talquetamab) (Experimental): Cohort B will enroll participants with multiple myeloma who have previously received >= 3 prior lines of therapy and have been exposed to T cell redirection therapies. Participants will receive talquetamab subcutaneously (SC) at a recommended Phase 2 dose (RP2D) selected after review of safety, efficacy, PK, and pharmacodynamic data from Part 1 and Part 2 of this study. All participants (ongoing and those who are in follow-up) will transition to OLE phase and will continue to receive the study treatment. Upon approval of amendment 19 and notification from the sponsor, participants will transition to the LTE and will continue to receive study treatment.
  Interventions: Drug: Talquetamab
- Part 3: Cohort C (Talquetamab) (Experimental): Cohort C will enroll participants with multiple myeloma who have previously received >= 3 prior lines of therapy and have not been exposed to T cell redirection therapies. Participants will receive talquetamab SC biweekly at a RP2D selected after review of safety, efficacy, PK, and pharmacodynamic data from Part 1 and Part 2 of this study. All participants (ongoing and those who are in follow-up) will transition to OLE phase and will continue to receive the study treatment. Upon approval of amendment 19 and notification from the sponsor, participants will transition to the LTE and will continue to receive study treatment.
  Interventions: Drug: Talquetamab
- Part 3: Cohort D (Talquetamab) (Experimental): Cohort D will enroll participants with multiple myeloma who have previously received >= 3 prior lines of therapy. Participants will receive talquetamab SC biweekly at a RP2D selected after review of safety, efficacy, PK, and pharmacodynamic data from Part 1 and Part 2 of this study. Participants in this cohort will receive tocilizumab prophylaxis for cytokine release syndrome (CRS) including all outpatient dosing. Participants will transition to OLE upon communication by the sponsor. Upon approval of amendment 19 and notification from the sponsor, participants will transition to the LTE and will continue to receive study treatment.
  Interventions: Drug: Talquetamab
- Part 3: Cohort E (Talquetamab) (Experimental): Cohort E will enroll participants with multiple myeloma who have previously received at least 1 proteasome inhibitor (PI), 1 immunomodulatory imide drug (IMiD), and 1 anti-cluster of differentiation 38 (CD38) monoclonal antibody.
  Participants will receive talquetamab SC biweekly at a RP2D selected after review of safety, efficacy, PK, and pharmacodynamic data from Part 1 and Part 2 of this study. Participants will receive tocilizumab prophylaxis for CRS with consolidated priming dose schedules as well as possible transition to outpatient priming dosing transition to OLE upon communication by the sponsor. Upon approval of amendment 19 and notification from the sponsor, participants will transition to the LTE and will continue to receive study treatment.
  Interventions: Drug: Talquetamab

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered SC until disease progression.
  Other Names: JNJ-64407564

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of talquetamab in participants with relapsed or refractory multiple myeloma at the recommended Phase 2 dose(s) (RP2Ds) (Part 3).

ELIGIBILITY:
Inclusion Criteria:

* Documented initial diagnosis of multiple myeloma according to international myeloma working group (IMWG) diagnostic criteria
* Part 3: Measurable disease cohort A, cohort B, cohort C and cohort D: multiple myeloma must be measurable by central laboratory assessment; Cohort E: Multiple myeloma must be measurable by local laboratory assessment
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2
* Women of childbearing potential must have a negative pregnancy test at screening and prior to the first dose of study drug using a highly sensitive pregnancy test either serum (beta human chorionic gonadotropin [hCG]) or urine
* Willing and able to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* Part 3 only: Cohort A and Cohort C only: exposed to a CAR-T or T cell redirection therapy at any time. Cohort B, Cohort D and Cohort E: T cell redirection therapy within 3 months
* Toxicities from previous anticancer therapies should have resolved to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy
* Received a cumulative dose of corticosteroids equivalent to >= 140 milligram (mg) of prednisone within the 14-day period before the first dose of study drug (does not include pretreatment medication)
* Stroke or seizure within 6 months prior to signing the informed consent form (ICF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years and 10 months
  ORR is defined as the proportion of participants who have a partial response (PR) or better according to the international myeloma working group (IMWG) criteria.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 2 years and 10 months
  DOR is defined as time from date of initial documentation of a response (PR or better) to date of first documented evidence of progressive disease (PD), per IMWG criteria, or death due to PD, whichever occurs first.
Very Good Partial Response (VGPR) or Better Rate | Up to 2 years and 10 months
  VGPR or better rate is defined as the percentage of patients who achieve a VGPR or better according to IMWG response criteria.
Complete Response (CR) or Better Rate | Up to 2 years and 10 months
  CR or better rate is defined as the percentage of patients who achieve CR or better according to IMWG response criteria.
Stringent Complete Response (sCR) Rate | Up to 2 years and 10 months
  sCR rate is defined as the percentage of patients who achieve sCR according to IMWG response criteria.
Time to Response (TTR) | Up to 2 years and 10 months
  TTR is defined as the time between date of first dose of study drug and the first efficacy evaluation that the participant has met all criteria for PR or better.
Progression-Free Survival (PFS) | Up to 2 years and 10 months
  PFS is defined as time from date of first dose of study drug to date of first documented PD, per IMWG criteria, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 2 years and 10 months
  OS is defined as the time from the date of first dose of study drug to the date of the participant's death.
Minimal Residual Disease (MRD) Negative Rate | Up to 2 years and 10 months
  MRD negativity rate is measured only for participants who achieve at least a CR but is reported based on all treated similar to the other response data.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 2 years and 10 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability | Up to 2 years and 10 months
  An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Number of Participants with AEs by Severity | Up to 2 years and 10 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE). Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to adverse event.
Number of Participants with Abnormalities in Clinical Laboratory Values | Up to 2 years and 10 months
  Number of participants with abnormalities in clinical laboratory values (such as hematology, serum chemistry and coagulation) will be reported.
Serum Concentration of Talquetamab | Up to 2 years and 10 months
  Serum samples will be analyzed to determine concentrations of talquetamab.
Number of Participants with Talquetamab Antibodies | Up to 2 years and 10 months
  Antibodies to talquetamab will be assessed to evaluate potential immunogenicity.
Change from Baseline in Health-Related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 item (EORTC QLQ-C30) | Baseline up to 2 years and 10 months
  The EORTC- QLQ-Core-30 includes 30 items that make up 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea/vomiting), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The recall period is 1 week ("past week") and responses are reported using a verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A higher score represents greater HRQoL, better functioning, and more (worse) symptoms.
Change from Baseline in HRQoL as Assessed by EuroQol Five Dimension Five Level Questionnaire (EQ-5D-5L) | Baseline up to 2 years and 10 months
  The EQ-5D-5L is a generic measure of health status. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). The scores for the 5 separate questions are categorical and cannot be analyzed as cardinal numbers.
Change from Baseline in HRQoL as Assessed by Patient Global Impression of Severity (PGIS) | Baseline up to 2 years and 10 months
  The PGIS is a single item that assesses severity of the participant's health state, on a 5-point verbal rating scale. Score ranges from 1 (None) to 5 (Very Severe).
Overall Response Rate (ORR) in Participants with High-risk Molecular Features | Up to 2 years and 10 months
  ORR in participants with high risk is defined as the overall response rate among the high risk molecular subgroups or other high-risk molecular subtypes.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (77):
- United States (14):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - Memorial Healthcare System, Hollywood, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Tennessee Oncology, Nashville, Tennessee
- Belgium (4):
  - UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
  - CHU de Liège - Domaine Universitaire du Sart Tilman, Liège
  - UCL - Saint Luc, Woluwe-Saint-Lambert
- China (7):
  - Peking University Third Hospital, Beijing
  - Sun Yat Sen University Cancer Center, Guangzhou
  - The 1St Affiliated Hospital of Medical College Zhejiang University, Hangzhou
  - First Affiliated Hospital SooChow University, Suzhou
  - Institute of Hematology & Blood Disease Hospital Chinese Academy of Medical Science, Tianjin
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- France (6):
  - CHU Henri Mondor, Créteil
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - C.H.U. Hotel Dieu - France, Nantes
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - Pôle IUC Oncopole CHU, Toulouse
- Germany (4):
  - Charite Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Muenster, Münster
  - Universitatsklinikum Wurzburg, Würzburg
- Israel (5):
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (13):
  - Kameda Medical Center, Chiba
  - Fukuoka University Hospital, Fukuoka
  - Ogaki Municipal Hospital, Gifu
  - Teine Keijinkai Hospital, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Kumamoto University Hospital, Kumamoto
  - Kurashiki Central Hospital, Kurashiki
  - National Hospital Organization Matsumoto Medical Center, Matsumoto
  - National Hospital Organization Okayama Medical Center, Okayama
  - Japanese Red Cross Osaka Hospital, Osaka
  - National Hospital Organization Hiroshima-Nishi Medical Center, Ōtake
  - Iwate Medical University Hospital, Shiwa-gun
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - UMCU, Utrecht
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut BadawczyOddz w Gliwicach, Gliwice
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- South Korea (6):
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (11):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Univ Vall D Hebron, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Virgen de La Arrixaca, Murcia
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Ito S, Kuroda Y, Sunami K, Matsue K, Imada K, Tamura H, Fujikawa E, Yamazaki H, Takamoto M, Pei L, Qin X, Masterson TJ, Campagna M, Vreys V, Lau BW, Takamatsu Y. Talquetamab in Japanese patients with relapsed/refractory multiple myeloma in the MonumenTAL-1 study. Int J Hematol. 2025 Dec 17. doi: 10.1007/s12185-025-04134-6. Online ahead of print. PMID 41405810
- [Derived] Einsele H, Moreau P, Bahlis N, Bhutani M, Vincent L, Karlin L, Perrot A, Goldschmidt H, van de Donk NWCJ, Ocio EM, Martinez Lopez J, Rodriguez-Otero P, Dytfeld D, Jakubowiak A, Schinke C, Besemer B, Anguille S, Manier S, Rasche L, Teipel R, Scheid C, Pawlyn C, Cavo M, Diels J, Ghilotti F, Lau BW, Renaud T, Orel O, Ong F, Ramos DF, Ammann E, Parekh T, Albrecht C, Weisel K, Mateos MV. Comparative Efficacy of Talquetamab vs. Real-World Physician's Choice of Treatment in Triple-Class-Exposed Relapsed/Refractory Multiple Myeloma: Updated Analyses of MonumenTAL-1 vs. LocoMMotion/MoMMent. Adv Ther. 2025 Nov 28. doi: 10.1007/s12325-025-03409-y. Online ahead of print. PMID 41313549
- [Derived] van de Donk NWCJ, Chari A, Martin T, Krishnan A, Rasche L, Ye JC, Popat R, Lipe B, Rodriguez C, Schinke C, Skerget S, Vishwamitra D, Verona R, Gong J, Singh I, Campagna M, Masterson T, Hilder B, Tolbert J, Renaud T, Smit MD, Heuck C, Mateos MV. Characterization and Management of Cytokine Release Syndrome From the MonumenTAL-1 Study of Talquetamab in Patients With Relapsed/Refractory Multiple Myeloma. Cancer Med. 2025 Oct;14(19):e71276. doi: 10.1002/cam4.71276. PMID 41036677
- [Derived] Schinke C, Rodriguez-Otero P, van de Donk NWCJ, Lipe B, Lavi N, Rasche L, Parekh S, Van Oekelen O, Vishwamitra D, Skerget S, Cortes-Selva D, Verona R, Hilder B, Masterson T, Campagna M, Khedkar S, Renaud T, Tolbert J, Kane C, Gray KS, Saber I, Heuck C, Chari A. Infections and parameters of humoral immunity with talquetamab in relapsed/refractory multiple myeloma in MonumenTAL-1. Blood Adv. 2025 Nov 25;9(22):5752-5762. doi: 10.1182/bloodadvances.2025016613. PMID 40864183
- [Derived] Schinke C, Touzeau C, Oriol A, Mateos MV, Stevens D, Rasche L, Qin X, Kato K, Bathija S, Katz EG, Gries KS, Campagna M, Masterson T, Hilder BW, Tolbert J, Renaud T, Heuck C, Tomlinson C, Moreau P, San-Miguel J, Rodriguez-Otero P, Chari A. Talquetamab improves patient-reported symptoms and health-related quality of life in relapsed or refractory multiple myeloma: Results from the phase 1/2 MonumenTAL-1 study. Cancer. 2025 Jul 15;131(14):e35927. doi: 10.1002/cncr.35927. PMID 40631904
- [Derived] Chari A, Touzeau C, Schinke C, Minnema MC, Berdeja JG, Oriol A, van de Donk NWCJ, Rodriguez-Otero P, Morillo D, Martinez-Chamorro C, Mateos MV, Costa LJ, Caers J, Rasche L, Krishnan A, Ye JC, Karlin L, Lipe B, Vishwamitra D, Skerget S, Verona R, Ma X, Qin X, Ludlage H, Campagna M, Masterson T, Hilder B, Tolbert J, Renaud T, Goldberg JD, Kane C, Heuck C, San-Miguel J, Moreau P. Safety and activity of talquetamab in patients with relapsed or refractory multiple myeloma (MonumenTAL-1): a multicentre, open-label, phase 1-2 study. Lancet Haematol. 2025 Apr;12(4):e269-e281. doi: 10.1016/S2352-3026(24)00385-5. Epub 2025 Mar 13. PMID 40090350
- [Derived] Catamero D, Ray C, Purcell K, Leahey S, Esler E, Rogers S, Hefner K, O'Rourke L, Gray K, Tolbert J, Renaud T, Patel S, Hannemann L, Shenoy S. Nursing Considerations for the Clinical Management of Adverse Events Associated with Talquetamab in Patients with Relapsed or Refractory Multiple Myeloma. Semin Oncol Nurs. 2024 Oct;40(5):151712. doi: 10.1016/j.soncn.2024.151712. Epub 2024 Aug 17. PMID 39155155
- [Derived] Einsele H, Moreau P, Bahlis N, Bhutani M, Vincent L, Karlin L, Perrot A, Goldschmidt H, van de Donk NWCJ, Ocio EM, Martinez-Lopez J, Rodriguez-Otero P, Dytfeld D, Diels J, Strulev V, Haddad I, Renaud T, Ammann E, Cabrieto J, Perualila N, Gan R, Zhang Y, Parekh T, Albrecht C, Weisel K, Mateos MV. Comparative Efficacy of Talquetamab vs. Current Treatments in the LocoMMotion and MoMMent Studies in Patients with Triple-Class-Exposed Relapsed/Refractory Multiple Myeloma. Adv Ther. 2024 Apr;41(4):1576-1593. doi: 10.1007/s12325-024-02797-x. Epub 2024 Feb 24. PMID 38402374
- See also: Dose Escalation Study of JNJ-64407564 in Participants With Relapsed or Refractory Multiple Myeloma — https://clinicaltrials.gov/ct2/show/NCT03399799